CLINICAL TRIAL: NCT04554849
Title: Demographic Characteristics and Psychosocial Health of Transgender People
Acronym: DyGeDem
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PI158
Record Dates: First submitted 2020-08-07; First posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-07

CONDITIONS: Gender Dysphoria
MeSH Terms: conditions — Gender Dysphoria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Gender dysphoria psychosocial health — Retrospective analysis of medical records

SUMMARY:
To study demographic characteristics of subjects referred to endocrine care for gender dysphoria and their psychosocial health

ELIGIBILITY:
Inclusion criteria - Person having received complete information on the organization of the research and willing to participate to research

Exclusion criteria:

- lack of data in the patients' records

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Subjects who met diagnostic criteria for gender dysphoria (International Classification of Diseases 11th Revision. https://icdwhoint. 2018) and were seen regularly in the outpatient clinic at our department of endocrinology
Study Population: Subjects who met diagnostic criteria for gender dysphoria (International Classification of Diseases 11th Revision. https://icdwhoint. 2018) and were seen regularly in the outpatient clinic at our department of endocrinology
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2020-07-24 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Retrospective analysis of medical records | 2004-2020
  Analysis of existing data

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided